CLINICAL TRIAL: NCT01182428
Title: A Clinical Evaluation of the XIENCE Everolimus Eluting Coronary Stent System in the Treatment of Women With de Novo Coronary Artery Lesions
Brief Title: XIENCE V: SPIRIT WOMEN Sub-study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-377 sub-study
Record Dates: First submitted 2010-07-13; First posted 2010-08-16 (Estimated); Results first posted 2012-07-13 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-07

CONDITIONS: Coronary Artery Stenosis; Coronary Arteriosclerosis; Coronary Artery Disease; Coronary Artery Restenosis; Total Coronary Occlusion; Stent Thrombosis; Vascular Disease; Myocardial Ischemia
Keywords: Stents; Angioplasty; Total coronary occlusions; Coronary restenosis; Stent thrombosis; Everolimus
MeSH Terms: conditions — Coronary Stenosis; Coronary Artery Disease; Coronary Restenosis; Vascular Diseases; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- XIENCE V® / XIENCE PRIME™ (Experimental)
  Interventions: Device: XIENCE V®/ XIENCE PRIME™
- CYPHER SELECT (Active Comparator)
  Interventions: Device: CYPHER SELECT

INTERVENTIONS:
Device: XIENCE V®/ XIENCE PRIME™ — Coronary artery placement of a XIENCE V®/ XIENCE PRIME™ Everolimus Eluting Stent System
  Arms: XIENCE V® / XIENCE PRIME™
Device: CYPHER SELECT — XIENCE V® / XIENCE PRIME™ to CYPHER SELECT in female patients with de novo coronary artery lesions
  Arms: CYPHER SELECT

SUMMARY:
The purpose of this Clinical Evaluation is the continued assessment of the XIENCE Everolimus Eluting Coronary Stent System (XIENCE V® and XIENCE PRIME™ EECSS) with the primary focus on clinical outcomes in the treatment of female patients with de novo coronary artery lesions, and the characterization of the female population undergoing stent implantation with a XIENCE stent.

DETAILED DESCRIPTION:
SPIRIT Women Randomized Sub-study is a prospective, single-blind, double arm, randomized multi-center sub-study comparing the XIENCE V® EECSS and XIENCE PRIME™ EESS to the CYPHER SELECT™ PLUS Sirolimus-eluting Coronary Stent in the treatment of female patients with coronary artery lesions.

The long term safety and efficacy of the XIENCE V EECSS have been demonstrated in the SPIRIT FIRST trial up to 5 years, the SPIRIT II trial up to 4 years, and in the SPIRIT III Randomized Control Trial (RCT) up to 3 years. In addition, these pre-approval studies have shown low rates of Target Vessel Failure and Major Adverse Cardiac Events (MACE) that were observed to plateau or gradually decline after about 1 year and were consistently lower than the comparator arm of each study. This benefit in MACE is sustained for up to 5 years and is also independent of the first year results.

The post approval SPIRIT V study demonstrated that the use of the XIENCE EECSS in complex lesions in a real-world population resulted in 1 year MACE, Stent Thrombosis and Target Lesion Revascularization rates that are comparable to those of the previously mentioned pre-approval studies which included patients with more restricted inclusion / exclusion criteria.

Therefore, based on existing data from these trials, Abbott Vascular has decided to discontinue further follow up in the SPIRIT Women study after 2 years.

ELIGIBILITY:
General Inclusion Criteria:

* Patient must be female.
* Patient must be at least 18 years of age.
* Patient is able to verbally confirm understanding of risks, benefits and treatment alternatives and she or her legally authorized representative provides written informed consent prior to any study related procedure, as approved by the appropriate Medical Ethics Committee of the respective clinical site.
* Patient must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or a reversible change in the electrocardiogram (ECG) consistent with ischemia).
* Patient must be an acceptable candidate for coronary artery bypass graft (CABG) surgery.
* Patient must agree to undergo all protocol-required follow-up examinations.
* Patients of childbearing potential must have had a negative pregnancy test within 7 days before treatment, and must not be nursing at the time of treatment.

Angiographic Inclusion Criteria:

* Patients' artery morphology and disease is suitable to be optimally treated with a maximum of 4 planned study stents.
* Target lesions must be de novo lesions (no prior stent implant, no prior brachytherapy).
* Target vessel reference diameter must be between 2.5 mm and 4.0 mm by visual estimate. The diameter range will be expanded to 2.25 mm when the 2.25 mm stent is available.
* Target lesion greater than or equal to 28 mm in length by visual estimate.

General Exclusion Criteria:

* Patient has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the clinical investigation plan, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year).
* Patient has a known hypersensitivity or contraindication to aspirin, either heparin or bivalirudin, both clopidogrel and ticlopidine, everolimus, cobalt, chromium, nickel, tungsten, acrylic and fluoro polymers or contrast sensitivity that cannot be adequately pre-medicated.
* Participation in another device or drug study or has completed the follow-up phase of another study within the last 30 days.
* Patient who is judged to have a lesion that prevents complete inflation of an angioplasty balloon.
* Patient has had a previous stent implant, either Bare Metal Stent (BMS) or Drug Eluting Stent (DES) within the target vessel(s)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2008-09; Primary Completion 2011-02 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Morice, Principal Investigator — Institut Cardiovasculaire Paris Sud (ICPS), Paris, France; Stephan Windecker, Principal Investigator — University Hospital Bern, Bern, Switzerland
Locations (25):
- Argentina (2):
  - Hosital Italiano de Buenos Aires - Cardiologia, Buenos Aires, Buenos Aires
  - Instituto Cardiovascular de Buenos Aires-ICBA, Buenos Aires
- Allgemeines Krankenhaus der Stadt Wien - Univ.Klinik f. Innere Medizin II, Vienna, Austria
- Heilig Hart Ziekenhuis Roeselare, Roeselare, Belgium
- Instituto de Cardiologia Dante Pazzanese Unidadae II Recepcao de Angioplastia, São Paulo, Brazil
- Rigshospitalet, Copenhagen, Denmark
- Institut Hospitalier Jacques Cartier Service d'Angiographie, Inst Cardiovasculaire Paris-Sud, Massy, France
- Germany (3):
  - Kardiologische Klinik Herz- und Diabeteszentrum, Bad Oeynhausen
  - Segebergerkliniken, Bad Segeberg
  - Technische Universität Dresden, Medizinische Klinik II - Kardiologie, Dresden
- Semmelweis University, Department of Cardiovascular Surgery, Budapest, Hungary
- Italy (5):
  - Centro Cardiologico Monzino, Milan
  - Clinico S.Ambrogio, GRUPPO OSPEDALIERO SAN DONATO, Milan
  - Azienda Policlinico di Modena U.O. Cardiologia, Ospedale di Modena, Modena
  - Ospedale Cisanello, Pisa
  - Istituto Clinico Humanitas, Rozzano
- Latvian Center of Cardiology, P. Stradina University Hospital, Riga, Latvia
- Netherlands (2):
  - AMC, Amsterdam
  - St. Antonius Ziekenhuis, Nieuwegein
- Haukeland university hospital, Bergen, Norway
- Institute of Cardiology, Warsaw, Poland
- Spain (2):
  - Hospital General de Alicante, Alicante
  - Hospital Universitari Germans Trias i Pujol, Barcelona
- Switzerland (2):
  - Inselspital Bern, Kardiologie, Bern
  - Cardiocentro Ticino, Lugano

REFERENCES:
- [Background] Morice MC. XIENCE V SPIRIT WOMEN clinical trial: characterization of the female population undergoing stent implantation. Womens Health (Lond). 2008 Sep;4(5):439-43. doi: 10.2217/17455057.4.5.439. PMID 19072483
- [Derived] Franzone A, Zaugg S, Piccolo R, Modena MG, Mikhail GW, Ferre JM, Strasser R, Grinfeld L, Heg D, Juni P, Windecker S, Morice MC. A randomized multicenter trial comparing the XIENCE everolimus eluting stent with the CYPHER sirolimus eluting stent in the treatment of female patients with de novo coronary artery lesions: The SPIRIT WOMEN study. PLoS One. 2017 Aug 10;12(8):e0182632. doi: 10.1371/journal.pone.0182632. eCollection 2017. PMID 28796809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between 30 Sept 2008 and 02 December 2009, from the general female interventional cardiology population who had been admitted for a PCI procedure.
Groups:
- XIENCE V® / XIENCE PRIME®: Subjects Randomized to XIENCE V®/XIENCE PRIME®. The number of participants at risk excludes subjects who are lost to follow up through 1 year without any event.
- CYPHER® SELECT: Subjects Randomized to CYPHER® SELECT. The number of participants at risk excludes subjects who are lost to follow up through 1 year without any event.
Period: Overall Study
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Started | 304 | 151
Completed | 293 | 150
Not Completed | 11 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 9 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT | Total
Number analyzed (Participants) | 304 | 151 | 455
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 105 | 42 | 147
  >=65 years | 199 | 109 | 308
Age Continuous [Mean (Standard Deviation); unit: years] | 68.37 (10.14) | 69.85 (10.54) | 68.86 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304 | 151 | 455
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 24 | 13 | 37
  Austria | 3 | 3 | 6
  Switzerland | 43 | 25 | 68
  Italy | 62 | 31 | 93
  France | 24 | 17 | 41
  Hungary | 41 | 12 | 53
  Argentina | 11 | 6 | 17
  Belgium | 6 | 4 | 10
  Brazil | 5 | 1 | 6
  Poland | 12 | 3 | 15
  Denmark | 16 | 5 | 21
  Germany | 26 | 13 | 39
  Latvia | 16 | 11 | 27
  Netherlands | 8 | 2 | 10
  Norway | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Adjudicated Composite Rate of All Death, All MI and Target Vessel Revascularization (TVR).
Description: This measure adds together all subjects who were determined by an expert panel to have died, had MI or had TVR as a result of their procedure.
Time Frame: at 1 year
Population: Based on Intent to Treat (ITT) population. The analysis population at follow-up visits may have changed due to early termination from the study by the patient or physician.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 293 | 150
Percentage of Participants | 21.5 [16.94 to 26.65] | 22 [15.65 to 29.49]

2. Secondary Outcome: Clinical Device Success
Description: Successful delivery and deployment of the study stent at the intended target lesion and successful withdrawal of the stent delivery system.
Time Frame: Intra-operative
Population: Based on Intent to Treat (ITT) population.
Measure: Number (95% Confidence Interval); unit: Percentage of evaluated lesions
Units Other Than Participants: Lesions
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 304 | 151
Number analyzed (Lesions) | 427 | 200
Percentage of evaluated lesions | 91.1 [87.99 to 93.63] | 93.5 [89.14 to 96.49]

3. Secondary Outcome: Clinical Procedure Success
Description: Successful delivery and deployment of the study stent or stents at the intended target lesion and successful withdrawal of the stent delivery system without adverse cardiac events.
Time Frame: Intra-operative
Population: Based on Intent to Treat (ITT) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 304 | 151
Percentage of Participants | 85.2 [80.70 to 88.99] | 84.1 [77.28 to 89.54]

4. Secondary Outcome: Adjudicated Stent Thrombosis (Definite, Probable)
Time Frame: < 1 day (Acute)
Population: Based on Intent to Treat (ITT) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 304 | 151
Percentage of Participants | 0.0 [0.0 to 1.21] | 0.0 [0.0 to 2.41]

5. Secondary Outcome: Adjudicated Stent Thrombosis (Definite, Probable)
Time Frame: 1 to 30 days (Sub-Acute)
Population: Based on Intent to Treat (ITT) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 304 | 151
Percentage of Participants | 0.0 [0.0 to 1.21] | 0.66 [0.02 to 3.63]

6. Secondary Outcome: Adjudicated Stent Thrombosis (Definite, Probable)
Time Frame: 30 days to 1 year (Late)
Population: Based on Intent to Treat (ITT) population. Population change based on follow up timeframe.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 287 | 144
Percentage of Participants | 0.0 [0.0 to 1.28] | 0.69 [0.02 to 3.81]

7. Secondary Outcome: Adjudicated Stent Thrombosis (Definite, Probable, Possible)
Time Frame: 30 days to 1 year (Late)
Population: Based on Intent to Treat (ITT) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 287 | 144
Percentage of Participants | 0.35 [0.01 to 1.93] | 1.39 [0.17 to 4.93]

8. Secondary Outcome: Adjudicated Composite Rate of Cardiac Death, MI Attributed to the Target Vessel and Clinically Indicated Target Lesion Revascularization (CI-TLR).
Time Frame: at 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 304 | 151
Percentage of Participants | 11.51 [8.15 to 15.65] | 13.25 [8.28 to 19.71]

9. Secondary Outcome: Adjudicated Composite Rate of Cardiac Death, MI Attributed to the Target Vessel and CI-TLR.
Time Frame: at 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 300 | 151
Percentage of Participants | 14.67 [10.86 to 19.18] | 14.57 [9.36 to 21.22]

10. Secondary Outcome: Adjudicated Composite Rate of Cardiac Death, MI Attributed to the Target Vessel and CI-TLR.
Time Frame: at 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 293 | 150
Percentage of Participants | 18.77 [14.47 to 23.72] | 18.67 [12.78 to 25.84]

11. Secondary Outcome: Adjudicated Composite Rate of All Death, All MI and Target Vessel Revascularization (TVR).
Time Frame: at 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 304 | 151
Percentage of Participants | 11.51 [8.15 to 15.65] | 13.25 [8.28 to 19.71]

12. Secondary Outcome: Adjudicated Composite Rate of All Death, All MI and Target Vessel Revascularization (TVR).
Time Frame: at 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 300 | 151
Percentage of Participants | 15.33 [11.45 to 19.92] | 15.23 [9.91 to 21.97]

13. Primary Outcome: In-stent Late Loss (LL) (Main Secondary Endpoint)
Description: In-stent Minimal Lumen Diameter (MLD)post-procedure - in-stent MLD at follow-up.
Time Frame: at 270 days
Population: The angiographic analysis population may be than the total population for the following reasons: Refusals, Death, Test Not Analyzable, Scheduling Problems, Medical Decisions, No study stent implanted, Patient Misunderstandings, Patient withdrawn by physician, Consent Withdrawal.
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Lesions
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 227 | 114
Number analyzed (Lesions) | 300 | 140
millimeters | 0.20 (0.38) | 0.12 (0.36)

14. Secondary Outcome: Adjudicated Composite Rate of All Death, All MI and All Revascularization (TLR/TVR/Non TVR).
Time Frame: at 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 304 | 151
Percentage of Participants | 12.17 [8.72 to 16.38] | 13.91 [8.82 to 20.47]

15. Secondary Outcome: Adjudicated Composite Rate of All Death, All MI and All Revascularization (TLR/TVR/Non TVR).
Time Frame: at 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 300 | 151
Percentage of Participants | 18.0 [13.82 to 22.82] | 17.88 [12.13 to 24.94]

16. Secondary Outcome: Adjudicated Composite Rate of All Death, All MI and All Revascularization (TLR/TVR/Non TVR).
Time Frame: at 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 293 | 151
Percentage of Participants | 27.99 [22.92 to 33.5] | 30 [22.8 to 38.01]

17. Secondary Outcome: Adjudicated Cardiac Death, Non-Cardiovascular Death, Vascular Death, Q-wave MI and Non Q-wave MI (Peri-Procedural, Unrelated to PCI).
Time Frame: at 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 304 | 151
Percentage of Participants | 11.51 [8.15 to 15.65] | 13.25 [8.28 to 19.71]

18. Secondary Outcome: Adjudicated Cardiac Death, Non-Cardiovascular Death, Vascular Death, Q-wave MI and Non Q-wave MI (Peri-Procedural, Unrelated to PCI).
Time Frame: at 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 300 | 151
Percentage of Participants | 12.67 [9.12 to 16.97] | 13.25 [8.28 to 19.71]

19. Secondary Outcome: Adjudicated Cardiac Death, Non-Cardiovascular Death, Vascular Death, Q-wave MI and Non Q-wave MI (Peri-Procedural, Unrelated to PCI).
Time Frame: at 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 293 | 150
Percentage of Participants | 13.99 [10.23 to 18.50] | 15.33 [9.98 to 22.11]

20. Secondary Outcome: In-segment Late Loss (LL)
Description: LL = Minimal Lumen Diameter (MLD) post-procedure minus MLD at follow-up
Time Frame: at 270 days
Population: The angiographic analysis population may be less than the total population for the following reasons: Refusals, Death, Test Not Analyzable, Scheduling Problems, Medical Decisions, No study stent implanted, Patient Misunderstandings, Patient withdrawn by physician, Consent Withdrawal.
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Lesions
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 227 | 114
Number analyzed (Lesions) | 299 | 140
millimeters | 0.10 (0.41) | 0.04 (0.37)

21. Secondary Outcome: In-stent Angiographic Binary Restenosis Rates
Description: Only a certain number of patients were required to have angiographic follow-up. Percent of subjects with a follow-up in-stent percent diameter stenosis of ≥ 50% per quantitative coronary angiography (QCA).
Time Frame: at 270 days
Population: The angiographic analysis population is less than the total population for the following reasons: Refusals, Death, Test Not Analyzable, Scheduling Problems, Medical Decisions, No study stent implanted, Patient Misunderstandings, Patient withdrawn by physician, Consent Withdrawal.
Measure: Number (95% Confidence Interval); unit: Percentage of Target Lesions
Units Other Than Participants: Target Lesion
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 227 | 114
Number analyzed (Target Lesion) | 314 | 148
Percentage of Target Lesions | 3.2 [1.54 to 5.78] | 0.7 [0.02 to 3.71]

22. Secondary Outcome: In-segment Angiographic Binary Restenosis Rates
Description: as for outcome 21
Time Frame: at 270 days
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: Percentage of target lesions
Units Other Than Participants: Target Lesions
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 227 | 114
Number analyzed (Target Lesions) | 305 | 144
Percentage of target lesions | 4.3 [2.29 to 7.18] | 2.1 [0.43 to 5.97]

23. Secondary Outcome: In-stent Percent Diameter Stenosis
Time Frame: at 270 days
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: % diameter stenosis
Units Other Than Participants: Target Lesions
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 227 | 114
Number analyzed (Target Lesions) | 314 | 148
% diameter stenosis | 15.77 (14.19) | 13.62 (11.10)

24. Secondary Outcome: In-segment Percent Diameter Stenosis
Time Frame: at 270 days
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: % diameter stenosis
Units Other Than Participants: Target Lesions
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 227 | 114
Number analyzed (Target Lesions) | 305 | 144
% diameter stenosis | 22.26 (13.45) | 20.14 (12.63)

25. Secondary Outcome: Adjudicated Revascularization (TLR/TVR/All Revascularizations)
Description: Composite of Target Lesion Revascularization (TLR), Target Vessel Revascularization (TVR), all revascularizations
Time Frame: at 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 304 | 151
Percentage of Participants | 0.66 [0.08 to 2.36] | 1.99 [0.41 to 5.7]

26. Secondary Outcome: Adjudicated Revascularization (TLR/TVR/All Revascularizations)
Description: Composite of Target Lesion Revascularization (TLR), Target Vessel Revascularization (TVR), all revascularizations
Time Frame: at 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 300 | 151
Percentage of Participants | 8.0 [5.19 to 11.67] | 5.96 [2.76 to 11.01]

27. Secondary Outcome: Adjudicated Revascularization (TLR/TVR/All Revascularizations)
Description: Composite of Target Lesion Revascularization (TLR), Target Vessel Revascularization (TVR), all revascularizations
Time Frame: at 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 293 | 150
Percentage of Participants | 18.09 [13.85 to 22.98] | 19.33 [13.35 to 26.57]

28. Secondary Outcome: Aneurysm
Description: All subjects with aneurysm of the target lesion up to the 270 day follow-up visit
Time Frame: at 270 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % of target lesions with aneurysm
Units Other Than Participants: Lesions
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 304 | 151
Number analyzed (Lesions) | 318 | 151
% of target lesions with aneurysm | 0.0 [0.0 to 1.15] | 0.0 [0.0 to 2.41]

29. Secondary Outcome: Thrombus
Description: All subjects with thrombus of the target lesion up to the 270 day follow-up visit
Time Frame: at 270 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of evaluated lesions
Units Other Than Participants: Lesions
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 304 | 151
Number analyzed (Lesions) | 317 | 151
Percentage of evaluated lesions | 0.3 [0.01 to 1.74] | 1.3 [0.16 to 4.70]

30. Secondary Outcome: Persisting Dissection
Description: All subjects with persisting dissection of the target lesion up to the 270 day follow-up visit
Time Frame: at 270 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of evaluated lesions
Units Other Than Participants: Lesions
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Number analyzed (Participants) | 304 | 151
Number analyzed (Lesions) | 306 | 145
Percentage of evaluated lesions | 0.0 [0.0 to 1.2] | 0.0 [0.0 to 2.51]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | XIENCE V® / XIENCE PRIME® | CYPHER® SELECT
Serious Adverse Events (participants affected / at risk) | 120/304 | 61/151
Other Adverse Events (participants affected / at risk) | 39/297 | 11/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | XIENCE V® / XIENCE PRIME® (N=304) | CYPHER® SELECT (N=151)
Anaemia (Blood and lymphatic system disorders) | 1/297 (1) | 4/149 (10)
Acute coronary syndrome (Cardiac disorders) | 0/297 (0) | 1/149 (1)
Acute myocardial infarction (Cardiac disorders) | 2/297 (2) | 0/149 (0)
Angina pectoris (Cardiac disorders) | 38/297 (44) | 8/149 (10)
Angina unstable (Cardiac disorders) | 8/297 (9) | 2/149 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 1/297 (1) | 0/149 (0)
Atrial fibrillation (Cardiac disorders) | 1/297 (1) | 1/149 (1)
Atrial flutter (Cardiac disorders) | 2/297 (3) | 0/149 (0)
Cardiac aneurysm (Cardiac disorders) | 1/297 (1) | 0/149 (0)
Ventricular tachycardia (Cardiac disorders) | 1/297 (1) | 0/149 (0)
Cardiac failure (Cardiac disorders) | 3/297 (3) | 2/149 (2)
Cardiac failure acute (Cardiac disorders) | 1/297 (1) | 1/149 (1)
Cardiac tamponade (Cardiac disorders) | 1/297 (1) | 0/149 (0)
Cardiogenic shock (Cardiac disorders) | 0/297 (0) | 1/149 (1)
Coronary artery disease (Cardiac disorders) | 1/297 (1) | 0/149 (0)
Coronary artery dissection (Cardiac disorders) | 1/297 (1) | 1/149 (1)
Coronary artery stenosis (Cardiac disorders) | 5/297 (5) | 6/149 (6)
Myocardial infarction (Cardiac disorders) | 5/297 (5) | 3/149 (3)
Myocardial ischaemia (Cardiac disorders) | 1/297 (1) | 1/149 (1)
Palpitations (Cardiac disorders) | 1/297 (1) | 1/149 (1)
Pericardial effusion (Cardiac disorders) | 1/297 (1) | 0/149 (0)
Tachycardia (Cardiac disorders) | 1/297 (1) | 0/149 (0)
Deafness (Ear and labyrinth disorders) | 0/297 (0) | 1/149 (1)
Vertigo positional (Ear and labyrinth disorders) | 0/297 (0) | 1/149 (1)
Diplopia (Eye disorders) | 1/297 (1) | 0/149 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1/297 (1) | 0/149 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1/297 (1) | 0/149 (0)
Gastric ulcer (Gastrointestinal disorders) | 1/297 (1) | 1/149 (1)
Haematochezia (Gastrointestinal disorders) | 1/297 (1) | 0/149 (0)
Ileus (Gastrointestinal disorders) | 0/297 (0) | 1/149 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1/297 (1) | 0/149 (0)
Melaena (Gastrointestinal disorders) | 0/297 (0) | 1/149 (1)
Periodontitis (Gastrointestinal disorders) | 1/297 (1) | 0/149 (0)
Asthenia (General disorders) | 1/297 (1) | 0/149 (0)
Catheter site haematoma (General disorders) | 5/297 (5) | 1/149 (1)
Catheter site haemorrhage (General disorders) | 1/297 (1) | 1/149 (1)
Chest discomfort (General disorders) | 2/297 (5) | 1/149 (1)
Non-cardiac chest pain (General disorders) | 1/297 (1) | 3/149 (3)
Cholecystitis (Hepatobiliary disorders) | 0/297 (0) | 1/149 (1)
Hypersensitivity (Immune system disorders) | 2/297 (2) | 0/149 (0)
Bronchitis (Infections and infestations) | 0/297 (0) | 1/149 (1)
Cystitis (Infections and infestations) | 0/297 (0) | 1/149 (1)
Diverticulitis (Infections and infestations) | 1/297 (1) | 0/149 (0)
Localised infection (Infections and infestations) | 1/297 (1) | 0/149 (0)
Pneumonia (Infections and infestations) | 2/297 (2) | 0/149 (0)
Urinary tract infection (Infections and infestations) | 0/297 (0) | 1/149 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1/297 (1) | 0/149 (0)
Concussion (Injury, poisoning and procedural complications) | 1/297 (1) | 0/149 (0)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1/297 (1) | 0/149 (0)
Device dislocation (Injury, poisoning and procedural complications) | 0/297 (0) | 1/149 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0/297 (0) | 1/149 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 2/297 (2) | 0/149 (0)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 1/297 (1) | 0/149 (0)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 5/297 (5) | 6/149 (6)
Nephropathy toxic (Injury, poisoning and procedural complications) | 1/297 (1) | 0/149 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1/297 (1) | 0/149 (0)
Reperfusion injury (Injury, poisoning and procedural complications) | 0/297 (0) | 1/149 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1/297 (1) | 0/149 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1/297 (1) | 0/149 (0)
Thrombosis in device (Injury, poisoning and procedural complications) | 0/297 (0) | 1/149 (1)
Biopsy breast (Investigations) | 1/297 (1) | 0/149 (0)
Blood creatine phosphokinase increased (Investigations) | 1/297 (1) | 0/149 (0)
Haemoglobin decreased (Investigations) | 1/297 (1) | 1/149 (1)
Troponin increased (Investigations) | 3/297 (3) | 0/149 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0/297 (0) | 1/149 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0/297 (0) | 1/149 (1)
Knee deformity (Musculoskeletal and connective tissue disorders) | 0/297 (0) | 1/149 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1/297 (1) | 0/149 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/297 (1) | 0/149 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/297 (0) | 1/149 (1)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/297 (1) | 0/149 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/297 (1) | 0/149 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/297 (1) | 0/149 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/297 (0) | 1/149 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/297 (1) | 0/149 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/297 (1) | 0/149 (0)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/297 (1) | 0/149 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/297 (1) | 0/149 (0)
Cerebral infarction (Nervous system disorders) | 1/297 (1) | 0/149 (0)
Dizziness (Nervous system disorders) | 1/297 (2) | 0/149 (0)
Headache (Nervous system disorders) | 2/297 (2) | 1/149 (1)
Hypoaesthesia (Nervous system disorders) | 0/297 (0) | 1/149 (1)
Paresis (Nervous system disorders) | 1/297 (1) | 0/149 (0)
Syncope (Nervous system disorders) | 1/297 (1) | 1/149 (1)
Transient ischaemic attack (Nervous system disorders) | 0/297 (0) | 2/149 (2)
Vascular dementia (Nervous system disorders) | 0/297 (0) | 1/149 (1)
Renal colic (Renal and urinary disorders) | 0/297 (0) | 1/149 (1)
Renal failure (Renal and urinary disorders) | 0/297 (0) | 1/149 (1)
Renal failure acute (Renal and urinary disorders) | 0/297 (0) | 1/149 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1/297 (1) | 0/149 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/297 (1) | 0/149 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4/297 (4) | 1/149 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0/297 (0) | 1/149 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0/297 (0) | 1/149 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/297 (0) | 1/149 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1/297 (1) | 0/149 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/297 (1) | 0/149 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1/297 (1) | 0/149 (0)
Arterial stent insertion (Surgical and medical procedures) | 0/297 (0) | 1/149 (1)
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 0/297 (0) | 1/149 (1)
Cataract operation (Surgical and medical procedures) | 0/297 (0) | 2/149 (2)
Coronary angioplasty (Surgical and medical procedures) | 0/297 (0) | 2/149 (2)
Coronary revascularisation (Surgical and medical procedures) | 1/297 (1) | 0/149 (0)
Hip arthroplasty (Surgical and medical procedures) | 0/297 (0) | 1/149 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 5/297 (5) | 2/149 (2)
Scar excision (Surgical and medical procedures) | 1/297 (1) | 0/149 (0)
Aortic aneurysm (Vascular disorders) | 1/297 (1) | 0/149 (0)
Arterial stenosis limb (Vascular disorders) | 0/297 (0) | 1/149 (1)
Duodenal ulcer haemorrhage (Vascular disorders) | 1/297 (1) | 0/149 (0)
Femoral arterial stenosis (Vascular disorders) | 1/297 (1) | 0/149 (0)
Gastric haemorrhage (Vascular disorders) | 1/297 (1) | 0/149 (0)
Gastrointestinal haemorrhage (Vascular disorders) | 3/297 (3) | 1/149 (1)
Hypertension (Vascular disorders) | 1/297 (1) | 0/149 (0)
Hypertensive crisis (Vascular disorders) | 0/297 (0) | 1/149 (2)
Intermittent claudication (Vascular disorders) | 2/297 (2) | 0/149 (0)
Lymphoedema (Vascular disorders) | 1/297 (1) | 0/149 (0)
Peripheral ischaemia (Vascular disorders) | 1/297 (1) | 0/149 (0)
Rectal haemorrhage (Vascular disorders) | 1/297 (1) | 0/149 (0)
Retroperitoneal hematoma (Vascular disorders) | 1/297 (1) | 0/149 (0)
Shock haemorrhagic (Vascular disorders) | 0/297 (0) | 1/149 (1)
Vascular pseudoaneurysm (Vascular disorders) | 5/297 (5) | 0/149 (0)
Cardiac enzymes increased (Investigations) | 2/297 (2) | 4/149 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XIENCE V® / XIENCE PRIME® (N=297) | CYPHER® SELECT (N=149)
Angina pectoris (Cardiac disorders) | 21 (22) | 4 (4)
Cardiac enzymes increased (Investigations) | 18 (18) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days